CLINICAL TRIAL: NCT02413346
Title: A Multi-Center Open-Label Evaluation of the Safety of Sarecycline Tablets in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC1403
Record Dates: First submitted 2015-04-02; First posted 2015-04-09 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — sarecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo/Sarecycline (Experimental): Participants received placebo-matching sarecyline in the double-blind lead-in study for up to 12 weeks; followed by, 1.5 milligram(mg)/kilogram(kg) sarecycline once daily (administered orally as 60 mg, 100 mg or 150 mg of sarecycline based on the participant's body weight) until adequate improvement in facial acne is obtained with re-initiation if acne recurs in this open-label study (Up to 40 weeks).
  Interventions: Drug: Sarecycline
- Sarecycline/Sarecycline (Experimental): Participants received sarecyline in the double-blind lead-in study for up to 12 weeks; followed by, 1.5 mg/kg sarecycline once daily (administered orally as 60 mg, 100 mg or 150 mg of sarecycline based on the participant's body weight) until adequate improvement in facial acne is obtained with re-initiation if acne recurs in this open-label study (Up to 40 weeks).
  Interventions: Drug: Sarecycline

INTERVENTIONS:
Drug: Sarecycline — Administered based on participant's body weight.

SUMMARY:
Open-label study will evaluate the safety of an approximate 1.5 mg/kg/day dose of oral sarecycline in the long-term treatment of participants with moderate to severe facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed participation in Phase 3 study of sarecycline (SC1401 or SC1402)
* Signed informed consent or assent form
* Body weight between 33 kg and 136 kg, inclusive
* Negative urine pregnancy test for females of childbearing potential
* Agrees to use effective method of contraception throughout study, if applicable.
* Able to fulfill protocol requirements, indicated willingness to participate in study and agrees to all study procedures by providing written informed consent/assent and authorization to disclose (personal health information)

Exclusion Criteria:

* Currently participating in another clinical study, unless it is a pharmacokinetic sarecycline study and participation approved by medical monitor; has received investigational medication (except sarecycline) within 30 days of enrollment.
* Discontinued participation in a Phase 3 study with sarecycline for any reason
* Had poor compliance wtih study requirements/study drug dosing in a Phase 3 study with sarecycline
* Is receiving/planning to receive any systemic acne medication, systemic retinoids, systemic corticosteroids or any androgen/anti-androgenic therapy (eg, testosterone, spironolactone)
* Is pregnant, lactating or planning a pregnancy during the study period
* Has a significant intercurrent illness (including clinically significant abnormality in clinical laboratory tests), psychiatric disorder, or other factors that, in the opinion of the Investigator or Medical Monitor, precludes participation in the study
* Is judged by the Investigator to be unsuitable for any reason

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Allergan, plc
Locations (56):
- United States (56):
  - Actavis Investigational Study Site #206, Mobile, Alabama
  - Actavis Investigational Study Site #236, Hot Springs, Arkansas
  - Actavis Investigational Study Site #245, Carlsbad, California
  - Actavis Investigational Study Site #129, Encino, California
  - Actavis Investigational Study Site #209, Fremont, California
  - Actavis Investigational Study Site #147, Sacramento, California
  - Actavis Investigational Study Site #150, San Diego, California
  - Actavis Investigational Study Site #125, San Diego, California
  - Actavis Investigational Study Site #204, San Diego, California
  - Actavis Investigational Study Site #222, Denver, Colorado
  - Actavis Investigational Study Site #148, Wheat Ridge, Colorado
  - Actavis Investigational Study Site #226, Clearwater, Florida
  - Actavis Investigational Study Site #238, Jupiter, Florida
  - Actavis Investigational Study Site #249, Miami, Florida
  - Actavis Investigational Study Site #145, Miami, Florida
  - Actavis Investigational Study Site #211, Miramar, Florida
  - Actavis Investigation Study Site # 140, North Miami Beach, Florida
  - Actavis Investigational Study Site #151, Orange, Florida
  - Actavis Investigational Study Site #203, Tampa, Florida
  - Actavis Investigational Study Site #242, Snellville, Georgia
  - Actavis Investigational Study Site #124, Boise, Idaho
  - Actavis Investigational Study Site #106, Chicago, Illinois
  - Actavis Investigational Study Site #113, South Bend, Indiana
  - Actavis Investigational Study Site #213, Louisville, Kentucky
  - Actavis Investigational Study Site #217, Rockville, Maryland
  - Actavis Investigational Study Site #251, Clarkston, Michigan
  - Actavis Investigational Study Site #235, Clinton Township, Michigan
  - Actavis Investigational Study Site #227, Fort Gratiot, Michigan
  - Actavis Investigational Study Site #111, Warren, Michigan
  - Actavis Investigational Study Site #221, Fridley, Minnesota
  - Actavis Investigational Study Site #231, Omaha, Nebraska
  - Actavis Investigational Study Site #146, New York, New York
  - Actavis Investigational Study Site #208, New York, New York
  - Actavis Investigational Study Site #240, Rochester, New York
  - Actavis Investigational Study Site #230, Stony Brook, New York
  - Actavis Investigational Study Site #229, Raleigh, North Carolina
  - Actavis Investigational Study Site #149, Gresham, Oregon
  - Actavis Investigational Study Site #257, Philadelphia, Pennsylvania
  - Actavis Investigational Study Site #225, Goodlettsville, Tennessee
  - Actavis Investigational Study Site #128, Knoxville, Tennessee
  - Actavis Investigational Study Site #216, Knoxville, Tennessee
  - Actavis Investigational Study Site #109, Nashville, Tennessee
  - Actavis Investigational Study Site #223, Arlington, Texas
  - Actavis Investigational Study Site #252, Arlington, Texas
  - Actavis Investigational Study Site #220, College Station, Texas
  - Actavis Investigational Study Site #104, Dallas, Texas
  - Actavis Investigational Study Site #142, Houston, Texas
  - Actavis Investigational Study Site #105, Houston, Texas
  - Actavis Investigational Study Site #201, Katy, Texas
  - Actavis Investigational Study Site #223, Pflugerville, Texas
  - Actavis Investigational Study Site #101, Plano, Texas
  - Actavis Investigational Study Site #207, San Antonio, Texas
  - Actavis Investigational Study Site #212, West Jordan, Utah
  - Actavis Investigational Study Site #244, Norfolk, Virginia
  - Actavis Investigational Study Site #144, Spokane, Washington
  - Actavis Investigational Study Site #233, Walla Walla, Washington

REFERENCES:
- [Derived] Pariser DM, Green LJ, Lain EL, Schmitz C, Chinigo AS, McNamee B, Berk DR. Safety and Tolerability of Sarecycline for the Treatment of Acne Vulgaris: Results from a Phase III, Multicenter, Open-Label Study and a Phase I Phototoxicity Study. J Clin Aesthet Dermatol. 2019 Nov;12(11):E53-E62. Epub 2019 Nov 1. PMID 32038757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Long-term safety study for participants who were treated for moderate to severe facial acne vulgaris in the double-blind studies SC1401 [NCT02320149] or SC1402 [NCT02322866].
Period: Overall Study
Arm/Group | Placebo/Sarecycline | Sarecycline/Sarecycline
Started | 236 | 247
Completed | 177 | 177
Not Completed | 59 | 70
Not completed — Adverse Event | 6 | 6
Not completed — Withdrawal by Subject | 30 | 40
Not completed — Lost to Follow-up | 17 | 21
Not completed — Protocol Violation | 2 | 0
Not completed — Other Miscellaneous Reasons | 4 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants among the screened population who were exposed to study treatment (sarecycline) in either the double-blind lead-in study or this open-label extension study.
Groups:
- Placebo/Sarecycline: Participants received placebo-matching sarecyline in the double-blind lead-in study for up to 12 weeks; followed by, 1.5 mg/kg sarecycline once daily (administered orally as 60 mg, 100 mg or 150 mg of sarecycline based on the participant's body weight) until adequate improvement in facial acne is obtained with re-initiation if acne recurs in this open-label study (Up to 40 weeks).
- Total: Total of all reporting groups
Arm/Group | Placebo/Sarecycline | Sarecycline/Sarecycline | Total
Number analyzed (Participants) | 236 | 247 | 483
Age, Customized [Number; unit: participants]
  ≥9 and <12 years | 2 | 3 | 5
  ≥12 and <18 years | 138 | 152 | 290
  ≥18 years | 96 | 92 | 188
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 125 | 247
  Male | 114 | 122 | 236

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. A TEAE is an AE that occurs after the first dose of study drug.
Time Frame: Up to 40 Weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo/Sarecycline | Sarecycline/Sarecycline
Number analyzed (Participants) | 236 | 247
participants | 94 | 94

ADVERSE EVENTS:
Time Frame: Signing of informed consent for this open-label study to end of study (Up to 40 Weeks)
Arm/Group | Placebo/Sarecycline | Sarecycline/Sarecycline
All-Cause Mortality (participants affected / at risk) | 0/236 | 0/247
Serious Adverse Events (participants affected / at risk) | 2/236 | 2/247
Other Adverse Events (participants affected / at risk) | 13/236 | 5/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sarecycline (N=236) | Sarecycline/Sarecycline (N=247)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sarecycline (N=236) | Sarecycline/Sarecycline (N=247)
Nasopharyngitis (Infections and infestations) | 13 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.